CLINICAL TRIAL: NCT01934569
Title: Evaluation Of The Effect Of PF-05089771 On The Metabolism Of Multiple Cytochrome P450 And OATP1B1 Transporter Substrates
Brief Title: Drug-Drug Interaction Study With PF-05089771
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B3291023
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
MeSH Terms: interventions — Pravastatin; Midazolam; Losartan; Omeprazole; Caffeine; PF-05089771

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active tratment (Experimental): Pravastatin, midazolam, losartan, omeprazole, caffeine single dose alone or in combination with PF-05089771
  Interventions: Drug: Pravastatin, midazolam, losartan, omeprazole, caffeine and PF-05089771

INTERVENTIONS:
Drug: Pravastatin, midazolam, losartan, omeprazole, caffeine and PF-05089771 — PF-05089771 450mg single dose and titration from 150mg BID to 450mg BID Pravastatin 10mg dingle dose, Midazolam 7.5mg single dose, Losartan 25mg single dose, Caffeine 100mg single dose, Omeprazole 20mg single dose

SUMMARY:
This study will test the potential for PF-05089771 to interact with a cocktail of drugs

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years;
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs);

Exclusion Criteria:

* Any condition possibly affecting drug absorption
* History of regular alcohol consumption
* Screening supine blood pressure >140 mm Hg (systolic) or >90 mm Hg (diastolic),
* Consumption of coffee, cola or other caffeine containing drinks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | 24h
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 24h
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Minimum Observed Plasma Trough Concentration (Cmin) | 24h
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 24h

SECONDARY OUTCOMES:
Change from Baseline in Lipid Parameters | 14 days
  Mean Total Cholesterol (TC), Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL), and Triglyceride blood concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291023&StudyName=Drug-Drug%20Interaction%20Study%20With%20PF-05089771%20